CLINICAL TRIAL: NCT05867212
Title: Implementation and Delivery of Cabotegravir Long Acting Injection for PrEP in a Community Pharmacy Setting.
Acronym: IDCaPP
Status: Completed | Type: Observational
Sponsor: Kelley-Ross & Associates, Inc. (Other)
Responsible Party: Principal Investigator, Elyse Tung, Director of Clinical Services, Kelley-Ross & Associates, Inc.
Other Study IDs: 001
Record Dates: First submitted 2023-04-24; First posted 2023-05-19 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections
Keywords: Cabotegravir; pharmacy; HIV PrEP; pre-exposure prophylaxis; long acting injection; Apretude
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Cabotegravir Injection [Apretude] — People who want to get the long acting injectable will have the option in participating in surveys after their visit and have their electronic health records reviewed.

SUMMARY:
The goal of this demonstration project or observational study is to evaluate the feasibility and acceptability of a pharmacist-managed cabotegravir long acting injectable for PrEP program in a community pharmacy setting.

The main question it aims to answer are:

* Is the program feasible and acceptable at the end of 1 year of operations?
* What are the facilitators and barriers of the program? Participants who want to start the FDA approved cabotegravir long acting injectable medication for PrEP will have the option participating in surveys and a review of their electronic health records. Medication will be administered based on FDA approved labeling guidelines and their PrEP care will be part of standard of care per CDC.

Pharmacists who want to provide the service to their patients will have the option of participating in surveys pre and post implementation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at the time of screening
* Weight ≥ 35 kg
* HIV-negative status
* Willing to provide informed consent and undergo all required study procedures.

Exclusion Criteria:

* Unknown or positive HIV status
* Coadministration of drugs that significantly decrease cabotegravir concentrations according to the FDA package insert.
* Any participants that do not meet criteria for management under CDTA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 subjects who meet all the inclusion criteria, none of the exclusion criteria, and provide informed consent will be enrolled as study participants
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-05-13 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of participants recruited in PrEP care | initiation
  Percentage of participants recruited into PrEP care at initiation
Percentage of participants retained in PrEP care | 1 year
  Percentage of participants retained in PrEP care at the end of 1 year
Adherence rate | 1 year
  Number of participants who adhered to target injection windows period by completing injection appointments versus the number of participants who missed their target injection window period by not completing injection appointments
Age | initiation
  age in years at study initiation
Percentage Sex assigned at birth | initiation
  Percentage of people who were assigned female at birth or assigned male at birth
Percentage of people with Gender identity | initiation
  Percentage of people with gender identity of male, female, trans male, trans female, genderqueer or gender nonconforming, different identity, prefer not to answer at initiation of study.
Percentage of people in a certain race | initiation
  Percentage of people who identify as American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Pacific Islander, White, other, or prefer not to answer) race at initiation of study.
Percentage of people who identify in a certain ethnicity | initiation
  Percentage of people who identify hispanic or latino, not hispanic or latino, prefer not to answer) ethnicity at initiation of study.
Percentage of people with Insurance | 1 year
  Percentage of people with Medicaid, Medicare, commercial insurance, or uninsured throughout the study.
Percentage of people who have housing | 1 year
  Percentage of people who have a steady place to live, a place to live today but worried about losing it in the future, or do not have a steady place to live at initiation of study.
Percentage of people who have a primary care provider | initiation of study
  Percentage of people who have a primary care provider relationship at initiation of study.
Percentage of people with more than 1 sexual partner | initiation
  Percentage of people with more than 1 sexual partner at initiation of study.
Percentage of people with HIV positive sexual partner | initiation
  Percentage of people who have one or more sexual partner who is HIV positive at initiation.
Percentage of people who have inconsistent condom use during sex | initiation
  Percentage of people who have inconsistent condom use during sex.
Percentage of people who use injection drugs | initiation
  Percentage of people who use injection drugs
Percentage of people who use HIV post exposure prophylaxis (PEP) in the last 12 months | initiation
  Percentage of people who use HIV post exposure prophylaxis (PEP) in the last 12 months at initiation
Percentage of people who have a history of sexually transmitted infection in the previous 6 months | initiation
  Percentage of people who use HIV post exposure prophylaxis (PEP) in the last 12 months at initiation
Percentage of people of certain background characteristics | initiation
  A baseline questionnaire will be used at initiation to collect background characteristics to determine percentage of people of a race, ethnicity, gender identity, sex assigned at birth, marital status, education level, employment status, annual income, and living situation.
Percentage of people with risk of acquiring HIV at initiation | 1 year
  A baseline questionnaire will be used at initiation to collection information on percentage of people who engage in sex, has sex with and partner who is living with HIV, has sex without a condom, been diagnosed with an STI in the last 6 months, have used HIV post-exposure prophylaxis in the lat 12 months,
Percentage of people who are acceptable to cabotegravir long acting injectable for PrEP | initiation
  A 27 item questionnaire that will be given at baseline that explores the reason a person would like to be on an injection for PrEP, reasons for not being able to make injection appointments, and rating their feelings around judgement for being on an injection.
Percentage of people feeling satisfied with cabotegravir long acting injectable for PrEP | 1 year
  A 7 item questionnaire will be given at every follow up appointment that explores the reason someone wants to stay on an injectable for PrEP, how comfortable they feel being on the injection, reasons for not being able to make injection appointments, and rating their feelings around judgement for being on an injection.
Percentage of people who discontinue long acting cabotegravir for PrEP for a particular reason | discontinuation
  A 2 item questionnaire will be given a discontinuation that explores why a person discontinues long acting cabotegravir and what their HIV prevention strategy will be moving forward.
Percentage of Pharmacist providers who have certain attitudes to providing long acting cabotegravir for PrEP | at initiation
  A 5 point questionnaire that explores a pharmacists reasons for providing long acting injectable cabotegravir for PrEP, reasons for being able to or not being able to provide the service.
Percentage of pharmacist providers who are acceptable to providing long acting cabotegravir for PrEP | 6 months
  A 6 item questionnaire that explores the reasons a pharmacist is able to or not able to provide the service

SECONDARY OUTCOMES:
Number of STI | 1 year
  number of chlamydia, syphilis, and gonorrhea infections detected during study
Number of HIV seroconversions | 1 year
  Number of HIV seroconversions detected during the study, reason for patient discontinuation, pharmacist provider and patient perspectives on barriers and facilitators.
Percentage of people who discontinue long acting cabotegravir for PrEP for a particular reason | 1 year
  A 2 item questionnaire will be given a discontinuation that explores why a person discontinues long acting cabotegravir and what their HIV prevention strategy will be moving forward.
Percentage of pharmacists who believe in certain barriers in providing the service | 1 year
  A 6 item questionnaire that explores the reasons a pharmacist cannot provide the service
Percentage of pharmacists who believe in certain facilitators in providing the service | 1 year
  A 6 item questionnaire that explores the reasons a pharmacist can provide the service
Percentage of patients who believe in certain facilitators for using the service | 1 year
  A 7 item questionnaire will be given at every follow up appointment that explores the reason someone can use the service.
Percentage of patients who believe in certain barriers for using the service | 1 year
  A 7 item questionnaire will be given at every follow up appointment that explores the reason someone cannot use the service.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kelley-Ross Pharmacy at the Polyclinic, Seattle, Washington
  - Kelley-Ross Capitol Hill Pharmacy, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No